CLINICAL TRIAL: NCT05137860
Title: Efficacy of the Use of Bortezomib for the Treatment of Relapsed Leukemia or Positive Minimal Residual Disease
Brief Title: Efficacy of the Use of Bortezomib for the Treatment of Relapsed Leukemia or Positive MRD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Christian Omar Ramos-Peñafiel, MD, PhD, Principal Investigator, Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGMDI/21/204/03/67
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse; Chemotherapeutic Toxicity; Minimal Residual Disease
Keywords: Acute lymphoblastic leukemia; Bortezomib; Relapse; Minimal Residual Disease; Toxicity
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual; Recurrence | interventions — Bortezomib

STUDY DESIGN:
Intervention Model Description: Clinical Randomized Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Group (No Intervention): Each patient will receive their standard chemotherapy treatment for patients with relapsed Acute Lymphoblastic Leukemia based on the HyperCVAD scheme for a period of 12 weeks. Each chemotherapy cycle will be monitored by the health team corresponding to the Hematology service and the principal investigator.
- Bortezomib Treatment Group (Experimental): Each patient will receive their standard chemotherapy treatment for patients with relapsed Acute Lymphoblastic Leukemia based on the HyperCVAD scheme in combination with Bortezomib for a period of 12 weeks. Each chemotherapy cycle will be monitored by the health team corresponding to the Hematology service and the principal investigator.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Combination of Bortezomib with Standard Chemotherapy scheme for acute lymphoblastic patients in relapse.
  Other Names: Intervention Group
  Arms: Bortezomib Treatment Group

SUMMARY:
Various drugs have been added to different treatment regimens in order to improve the response rate in patients with Acute Lymphoblastic Leukemia, however, it has been shown that adding Bortezomib to the relapsing regimen improves the proportion of second complete remissions without increasing chemotherapy toxicity. Therefore, proteasome inhibitors can drastically modify the prognosis of patients, since their synergy with drugs such as steroids has positioned them as an attractive strategy.

DETAILED DESCRIPTION:
Mortality associated with leukemia has decreased due to the use of various chemotherapy combinations, the addition of new agents, or the chemical modification of existing drugs. Despite advances in treatment, the prognosis in the adult population continues to be unfavorable. About 25% of the patients will be refractory to the first treatment regimen and the rest will have a disease-free survival below 40%. The chemotherapy intensity reduction strategy based on risk stratification according to Minimal Residual Disease (MRD) is a strategy used by various pediatric centers in order to detect patients at high risk of relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmatory diagnosis of Acute Lymphoblastic Leukemia relapsed to bone marrow described with more than 5% blasts in bone marrow at any stage of treatment or positivity of minimal residual disease at any stage of treatment.
* Patients who have signed their informed consent from the institution for hospitalization, and accepted the performance of the bone marrow study, and the administration of chemotherapy.

Exclusion Criteria:

* Patients with a diagnosis of phenotypic leukemia or bilinear leukemia
* Patients treated only with palliative regimen or transfusion support
* Patients without the administration of prophylaxis to the central nervous system by intrathecal chemotherapy
* Patients with lymphoblastic leukemia with a positive Philadelphia chromosome
* Patients with severe comorbidities may put treatment therapy at risk.
* Patient with a history of cardiac toxicity or arrhythmias associated with treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-12-22 (Estimated); Study Completion 2023-06-23 (Estimated)

PRIMARY OUTCOMES:
Survival Outcome | 3 months
  The event in which patient is discharge from Hospital stay.
Hospital stay | 3 months
  Time in which patients stay in the Hospital before discharge
Leukocytes count | 3 months
  Number of leukocytes found in peripheral blood at the end of each chemotherapy cycle
Platelets count | 3 months
  Number of platelets found in peripheral blood at the end of each chemotherapy cycle
Date of Remission | 3 month
  Time in which the patient completes remission

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Martinez Tovar, PhD, Study Director — Hospital General de Mexico
Locations (1):
- Hospital General de México "Dr. Eduardo Liceaga", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
All participants and their information will be managed by intern investigators and will be kept secure for personal data protection according to Mexican laws.

REFERENCES:
- [Background] Burton JD, Bamford RN, Peters C, Grant AJ, Kurys G, Goldman CK, Brennan J, Roessler E, Waldmann TA. A lymphokine, provisionally designated interleukin T and produced by a human adult T-cell leukemia line, stimulates T-cell proliferation and the induction of lymphokine-activated killer cells. Proc Natl Acad Sci U S A. 1994 May 24;91(11):4935-9. doi: 10.1073/pnas.91.11.4935. PMID 8197160
- [Result] Bertaina A, Vinti L, Strocchio L, Gaspari S, Caruso R, Algeri M, Coletti V, Gurnari C, Romano M, Cefalo MG, Girardi K, Trevisan V, Bertaina V, Merli P, Locatelli F. The combination of bortezomib with chemotherapy to treat relapsed/refractory acute lymphoblastic leukaemia of childhood. Br J Haematol. 2017 Feb;176(4):629-636. doi: 10.1111/bjh.14505. Epub 2017 Jan 24. PMID 28116786
- [Result] Horton TM, Whitlock JA, Lu X, O'Brien MM, Borowitz MJ, Devidas M, Raetz EA, Brown PA, Carroll WL, Hunger SP. Bortezomib reinduction chemotherapy in high-risk ALL in first relapse: a report from the Children's Oncology Group. Br J Haematol. 2019 Jul;186(2):274-285. doi: 10.1111/bjh.15919. Epub 2019 Apr 7. PMID 30957229